CLINICAL TRIAL: NCT03770689
Title: A Multicenter Study With an Open-label Phase Ib Part Followed by a Randomized, Placebo-controlled, Double-blind, Phase II Part to Evaluate Efficacy, Safety, Tolerability, and Pharmacokinetics of the DNA-PK Inhibitor Peposertib (M3814) in Combination With Capecitabine and RT in Participants With Locally Advanced Rectal Cancer
Brief Title: Study of Peposertib in Combination With Capecitabine and RT in Rectal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MS100036_0020; 2018-002275-18 (EudraCT Number)
Record Dates: First submitted 2018-12-07; First posted 2018-12-10 (Actual); Results first posted 2022-07-07 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Locally Advanced Rectal Cancer
Keywords: DNA-PK inhibitor; Peposertib; capecitabine
MeSH Terms: interventions — peposertib; Capecitabine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Peposertib 50 mg + RT + Capecitabine (Experimental): Participants received peposertib 50 milligram (mg) once daily in combination with capecitabine 825 milligram per square meter (mg/m^2) twice daily 5 days per week and radiotherapy (RT) of 50 to 50.4 Gray (Gy) to the tumor area and 45 Gy to the electively irradiated tissues in 25 to 28 fractions up to 5.5 weeks treatment period.
  Interventions: Drug: Peposertib 50 mg; Drug: Capecitabine; Radiation: Radiotherapy (RT)
- Peposertib 100 mg + RT + Capecitabine (Experimental): Participants received peposertib 100 mg once daily in combination with capecitabine 825 mg/m^2 twice daily 5 days per week and RT of 50 to 50.4 Gy to the tumor area and 45 Gy to the electively irradiated tissues in 25 to 28 fractions up to 5.5 weeks treatment period.
  Interventions: Drug: Peposertib 100 mg; Drug: Capecitabine; Radiation: Radiotherapy (RT)
- Peposertib 150 mg + RT + Capecitabine (Experimental): Participants received peposertib 150 mg once daily in combination with capecitabine 825 mg/m^2 twice daily 5 days per week and RT of 50 to 50.4 Gy to the tumor area and 45 Gy to the electively irradiated tissues in 25 to 28 fractions up to 5.5 weeks treatment period.
  Interventions: Drug: Peposertib 150 mg; Drug: Capecitabine; Radiation: Radiotherapy (RT)
- Peposertib 250 mg + RT + Capecitabine (Experimental): Participants received peposertib 250 mg once daily in combination with capecitabine 825 mg/m^2 twice daily 5 days per week and RT of 50 to 50.4 Gy to the tumor area and 45 Gy to the electively irradiated tissues in 25 to 28 fractions up to 5.5 weeks treatment period.
  Interventions: Drug: Peposertib 250 mg; Drug: Capecitabine; Radiation: Radiotherapy (RT)

INTERVENTIONS:
Drug: Peposertib 50 mg — Participants received peposertib 50 milligram (mg) once daily 5 days per week up to 5.5 weeks.
  Other Names: M3814; MSC2490484A
  Arms: Peposertib 50 mg + RT + Capecitabine
Drug: Peposertib 100 mg — Participants received peposertib 100 mg once daily 5 days per week up to 5.5 weeks.
  Arms: Peposertib 100 mg + RT + Capecitabine
Drug: Peposertib 150 mg — Participants received peposertib 150 mg once daily 5 days per week up to 5.5 weeks.
  Arms: Peposertib 150 mg + RT + Capecitabine
Drug: Peposertib 250 mg — Participants received peposertib 250 mg once daily 5 days per week up to 5.5 weeks.
  Arms: Peposertib 250 mg + RT + Capecitabine
Drug: Capecitabine — Participants received capecitabine at a dose of 825 milligram per square meter (mg/m^2) twice daily 5 days per week up to 5.5 weeks.
Radiation: Radiotherapy (RT) — Participants received RT 50 to 50.4 Gray (Gy) to the tumor area and 45 Gy to the electively irradiated tissues in 25 to 28 fractions up to 5.5 weeks.

SUMMARY:
The main purpose of the study was to define maximum tolerated dose (MTD), recommended Phase II dose (RP2D) safety and tolerability of Peposertib in combination with capecitabine and radiotherapy (RT).

ELIGIBILITY:
Inclusion Criteria:

* Participants who have an Eastern Cooperative Oncology Group Performance Status less than or equals to (<=) 1
* Participants who have histologically confirmed and localized resectable rectal cancer (Stage 3)
* Participants who received induction chemotherapy are allowed to be enrolled to this study except this induction is resulting in clinical complete response (cCR) or tumor progression
* Participants who have lower edge of the tumor located in rectum
* Adequate hematological, hepatic and renal function as defined in the protocol
* Male participants if they agree to the following during the study intervention period and for at least 12 weeks after the last dose of study intervention
* Female participants are eligible if not pregnant or breastfeeding
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Participants with history of any other significant medical disease or psychiatric conditions that might in the assessment of the Investigator preclude safe participation in the study
* Participants with history of difficulty swallowing, malabsorption, or other chronic gastrointestinal disease or conditions that may hamper compliance and/or absorption of the study intervention
* Unstable cardiovascular function within 6 months prior to enrollment
* Hypertension uncontrolled by medication (ie, systolic blood pressure >= 150 millimeter of mercury (mmHg) and diastolic blood pressure >= 90 mmHg)
* Participants with history of other malignant disease within the past 5 years, other than successfully treated basal carcinoma of the skin or carcinoma in situ of the cervix
* Participants with known human immunodeficiency virus positivity, known active hepatitis (for example, hepatitis B virus or hepatitis C virus), current alcohol abuse, or cirrhosis
* Participants with ongoing active infection or treatment with a live attenuated vaccine within 4 weeks of dosing
* Participants with concomitant use of H2-blocker or proton pump inhibitors (PPIs) (or unable to stop at least 5 days prior to the first treatment). Note that calcium carbonate is acceptable
* Participation in any interventional clinical study within 28 days prior to Screening or during participation in this study
* Other protocol defined exclusion criteria could apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2021-06-21 (Actual); Study Completion 2022-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (14):
- United States (10):
  - University of Colorado Cancer Center, Aurora, Colorado
  - Yale University - Pediatric Respiratory Medicine, New Haven, Connecticut
  - Northwell Health, Inc, Great Neck, New York
  - Memorial Sloan-Kettering Cancer Center (MSKCC) - New York, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Ohio State University Clinical Trials Management Office - Ohio State CTMO Parent, Columbus, Ohio
  - University of Toledo Medical Center - Hematology/Oncology, Toledo, Ohio
  - Med. Univ. of South Carolina, Charleston, South Carolina
  - Greenville Hospital System University Medical Center (ITOR), Greenville, South Carolina
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Spain (4):
  - Hospital Universitari Vall d'Hebron - Dept of Oncology, Barcelona
  - Hospital Universitario 12 de Octubre - Servicio de Oncologia, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital Clinico Universitario de Valencia - Servicio de Hematologia y Oncologia Medica, Valencia

IPD SHARING:
Plan to Share IPD: No
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and the European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website bit.ly/IPD21

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS100036_0020
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html
- See also: DDRiver website — http://www.DDRiver-trials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was planned to be conducted in two phases: Phase Ib and Phase II. Phase II of the study was never initiated due to early discontinuation as per sponsor's decision.
Groups:
- Peposertib 50 mg + RT + Capecitabine:: Participants received peposertib 50 milligram (mg) once daily in combination with capecitabine 825 milligram per square meter (mg/m^2) twice daily 5 days per week and radiotherapy (RT) of 50 to 50.4 Gray (Gy) to the tumor area and 45 Gy to the electively irradiated tissues in 25 to 28 fractions up to 5.5 weeks treatment period.
- Peposertib 100 mg + RT + Capecitabine:: Participants received peposertib 100 mg once daily in combination with capecitabine 825 mg/m^2 twice daily 5 days per week and RT of 50 to 50.4 Gy to the tumor area and 45 Gy to the electively irradiated tissues in 25 to 28 fractions up to 5.5 weeks treatment period.
- Peposertib 150 mg + RT + Capecitabine:: Participants received peposertib 150 mg once daily in combination with capecitabine 825 mg/m^2 twice daily 5 days per week and RT of 50 to 50.4 Gy to the tumor area and 45 Gy to the electively irradiated tissues in 25 to 28 fractions up to 5.5 weeks treatment period.
- Peposertib 250 mg + RT + Capecitabine:: Participants received peposertib 250 mg once daily in combination with capecitabine 825 mg/m^2 twice daily 5 days per week and RT of 50 to 50.4 Gy to the tumor area and 45 Gy to the electively irradiated tissues in 25 to 28 fractions up to 5.5 weeks treatment period.
Period: Overall Study
Arm/Group | Peposertib 50 mg + RT + Capecitabine: | Peposertib 100 mg + RT + Capecitabine: | Peposertib 150 mg + RT + Capecitabine: | Peposertib 250 mg + RT + Capecitabine:
Started | 1 | 6 | 6 | 6
Pharmacokinetic Analysis Set | 1 (Number of participants analyzed in 50 mg group for PK outcome is different than PK analysis set. Because 1 participant from peposertib 100 mg took peposertib 50 mg from Fraction Day (FD) 1 through FD 10. PK results for this participant was summarized by actual dose received (50 mg) whereas non-PK results are summarized by planned dose (100 mg). Number of participants analyzed for 50 mg dose level in PK outputs that is 2 was therefore higher than non-PK outputs that is 1.) | 6 (Number of participants analyzed in 100 mg group for PK outcome is different than PK analysis set. Because 1 participant from peposertib 100 mg took peposertib 50 mg from Fraction Day (FD) 1 through FD 10. PK results for this participant was summarized by actual dose received (50 mg) whereas non-PK results are summarized by planned dose (100 mg). Number of participants analyzed for 100 mg dose level in PK outputs that is 5 was therefore lesser than non-PK outputs that is 6.) | 6 | 6
Full Analysis Set (FAS) | 1 | 6 | 6 | 6
Safety Analysis Set (SAF) | 1 | 6 | 6 | 6
Completed | 1 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety (SAF) analysis set included all participants who received at least 1 dose of study intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Peposertib 50 mg + RT + Capecitabine: | Peposertib 100 mg + RT + Capecitabine: | Peposertib 150 mg + RT + Capecitabine: | Peposertib 250 mg + RT + Capecitabine: | Total
Number analyzed (Participants) | 1 | 6 | 6 | 6 | 19
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60 | 60 (15.0) | 55 (8.9) | 58 (11.2) | 58 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 2 | 3 | 8
  Male | 1 | 3 | 4 | 3 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 1 | 6 | 6 | 5 | 18
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 1 | 6 | 6 | 6 | 19
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Dose Limiting Toxicity (DLT) Confirmed by Safety Monitoring Committee (SMC)
Description: DLT is defined as any of following treatment emergent adverse events (TEAEs) considered possibly related to study treatment by Investigator and/or Sponsor up to completion of assigned chemoradiotherapy treatment. DLT were based on SMC: Adverse drug reaction that, in the opinion of SMC, is of potential clinical significance such that further dose escalation would expose participants to unacceptable risk; Any occurrence of drug-induced liver injury meeting the Hy's law criteria; Any Grade 3 toxicity excluding diarrhea, neutropenia lasting for ≤ 5 days, nausea & vomiting, Grade 3 thrombocytopenia without bleeding; Grade ≥ 4 AEs at least possibly related to study drug, irrespective of duration, excluding: Isolated Grade 4 lymphocytopenia without clinical symptoms; Neutropenia lasting for ≤ 5 days and not associated with fever; Any toxicity related to study drug that causes participant to receive > 80% of planned peposertib, capecitabine or RT dose.
Time Frame: Time from first study intervention up to 19 weeks (including 5.5 weeks of treatment and 13.5 weeks of short term safety follow-up period)
Population: Dose escalation (DE) analysis set included all participants treated in dose escalation cohorts, who received at least 80% of peposertib, 50% of capecitabine, and 80% of RT planned dose and complete DLT period (5 or 5.5 weeks after start of treatment or for the entire duration of treatment). DE set also included participants treated in dose escalation cohorts who experience a DLT during DLT period regardless of the amount of each study intervention received/completion of the DLT period.
Measure: Count of Participants; unit: Participants
Arm/Group | Peposertib 50 mg + RT + Capecitabine: | Peposertib 100 mg + RT + Capecitabine: | Peposertib 150 mg + RT + Capecitabine: | Peposertib 250 mg + RT + Capecitabine:
Number analyzed (Participants) | 1 | 5 | 6 | 6
Participants | 0 | 1 | 1 | 3

2. Secondary Outcome: Number of Participants Wtih Treatment Emergent Adverse Events (TEAEs) and Treatment-Related TEAEs According to National Cancer Institute Common Terminology Criteria of Adverse Events (NCI-CTCAE) Version 5.0
Description: Adverse event (AE) is any untoward medical occurrence in participant administered pharmaceutical product, regardless of causal relationship with this treatment. Therefore, an AE can be any unfavorable & unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with use of a medicinal product, regardless if it is considered related to medicinal product. Serious AE: an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. TEAE: AE with onset after start of treatment or with onset date before the treatment start date but worsening after treatment start date. TEAEs included both serious and non-serious TEAEs. Treatment-related TEAEs: reasonably related to study intervention. Number of participants with TEAEs and treatment related TEAEs were reported.
Time Frame: Time from first study intervention up to long term safety follow-up period (Up to Month 35)
Population: SAF analysis set included all participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Peposertib 50 mg + RT + Capecitabine: | Peposertib 100 mg + RT + Capecitabine: | Peposertib 150 mg + RT + Capecitabine: | Peposertib 250 mg + RT + Capecitabine:
Number analyzed (Participants) | 1 | 6 | 6 | 6
Participants
  Participants with TEAEs | 1 | 6 | 6 | 6
  Participants with Treatment-Related TEAEs | 1 | 6 | 6 | 6

3. Secondary Outcome: Number of Participants With Abnormalities [Grade Greater Than or Equals to (>=) 3] in Laboratory Test Values
Description: The laboratory measurements included hematology and biochemistry values were graded with National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0 toxicity grades (where Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 = life threatening and Grade 5 = death). Number of participants with abnormalities Grade >= 3 in laboratory test values were reported.
Time Frame: Time from first study intervention up to long term safety follow-up period (Up to Month 35)
Population: SAF analysis set included all participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Peposertib 50 mg + RT + Capecitabine: | Peposertib 100 mg + RT + Capecitabine: | Peposertib 150 mg + RT + Capecitabine: | Peposertib 250 mg + RT + Capecitabine:
Number analyzed (Participants) | 1 | 6 | 6 | 6
Participants | 1 | 6 | 6 | 6

4. Secondary Outcome: Number of Participants With Markedly Abnormal Vital Sign Measurements
Description: Vital sign assessments included assessments of heart rate, diastolic blood pressure, systolic blood pressure, respiratory rate and temperature. Number of participants with markedly abnormal vital sign measurements were reported.
Time Frame: Time from first study intervention up to long term safety follow-up period (Up to Month 35)
Population: SAF analysis set included all participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Peposertib 50 mg + RT + Capecitabine: | Peposertib 100 mg + RT + Capecitabine: | Peposertib 150 mg + RT + Capecitabine: | Peposertib 250 mg + RT + Capecitabine:
Number analyzed (Participants) | 1 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Electrocardiogram (ECG) Findings
Description: Electrocardiograms (ECG) was obtained after the participant has been in a semi-supine position for at least 5 min. ECG parameters included heart rate, PQ/PR duration, QRS and QT duration, QT Interval. Clinical significance was determined by the investigator. Number of participants with clinically significant abnormalities in 12-lead ECG were reported.
Time Frame: Time from first study intervention up to long term safety follow-up period (Up to Month 35)
Population: SAF analysis set included all participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Peposertib 50 mg + RT + Capecitabine: | Peposertib 100 mg + RT + Capecitabine: | Peposertib 150 mg + RT + Capecitabine: | Peposertib 250 mg + RT + Capecitabine:
Number analyzed (Participants) | 1 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0

6. Secondary Outcome: Percentage of Participants With Composite Pathological Complete Response (pCR)/ Clinical Complete Response (cCR)
Description: pCR: It is defined as absence of viable tumor cells in the primary tumor and lymph nodes. Participants considered to have a pCR if they undergo surgery and no residual cancer is found on histological examination of removed specimen. cCR: Participants are considered to have a cCR if: 1) Absence of any residual tumor in primary site and draining lymph nodes on imaging with magnetic resonance imaging; 2) No visible lesion at endoscopy except a flat scar, telangiectasia, and/or whitening of mucosa; 3) Absence of any palpable tumor or irregularity on digital rectal examination (DRE) and endoscopic ultrasonography (EUS); 4) If a biopsy is taken, it must be negative. Participants are considered as responders to composite endpoint pCR/cCR if participant had surgery and had pCR; participant did not undergo surgery but had cCR. Number of participants with composite pathological complete response (pCR)/ clinical complete response (cCR) were reported.
Time Frame: At Week 15
Population: Full analysis set (FAS) include all participants who are enrolled in the study and received at least 1 dose of study intervention.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Peposertib 50 mg + RT + Capecitabine: | Peposertib 100 mg + RT + Capecitabine: | Peposertib 150 mg + RT + Capecitabine: | Peposertib 250 mg + RT + Capecitabine:
Number analyzed (Participants) | 1 | 6 | 6 | 6
percentage of participants | 0.0 [0.0 to 97.5] | 16.7 [0.4 to 64.1] | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 45.9]

7. Secondary Outcome: Disease-free Survival
Description: Disease-free Survival time, defined as the time from first treatment day to the date of the first documentation of objective progressive disease or death due to any cause, whichever occurs first. Median disease-free survival time was estimated according to Kaplan-Meier method.
Time Frame: Time from first study intervention up to approximately 35 months
Population: FAS include all participants who are enrolled in the study and received at least 1 dose of study intervention. As per the planned analysis, Kaplan-Meier estimates were planned to be presented as overall, together with a summary of associated statistics for this outcome measure.
Measure: Median (Full Range); unit: Months
Groups:
- Overall Participants: Participants received peposertib 50 mg, 100 mg, 150 mg and 250 mg in their respective cohort once daily in combination with capecitabine 825 milligram per square meter (mg/m^2) twice daily 5 days per week and radiotherapy (RT) of 50 to 50.4 Gray (Gy) to the tumor area and 45 Gy to the electively irradiated tissues in 25 to 28 fractions up to 5.5 weeks treatment period.
Arm/Group | Overall Participants
Number analyzed (Participants) | 19
Months | 21.2 [0.0 to 23.5]

8. Secondary Outcome: Percentage of Participants With Pathological Complete Response (pCR)
Description: pCR is defined as the absence of viable tumor cells in the primary tumor and lymph nodes. Participants are considered to have a pCR if they undergo surgery and no residual cancer is found on histological examination of the removed specimen.
Time Frame: At Week 15
Population: FAS include all participants who are enrolled in the study and received at least 1 dose of study intervention.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Peposertib 50 mg + RT + Capecitabine: | Peposertib 100 mg + RT + Capecitabine: | Peposertib 150 mg + RT + Capecitabine: | Peposertib 250 mg + RT + Capecitabine:
Number analyzed (Participants) | 1 | 6 | 6 | 6
percentage of participants | 0.0 [0.0 to 97.5] | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 45.9]

9. Secondary Outcome: Percentage of Participants With Clinical Complete Response (cCR)
Description: cCR: It is defined as participants considered to have a cCR if: 1) Absence of any residual tumor in the primary site and draining lymph nodes on imaging with magnetic resonance; 2) No visible lesion at endoscopy except a flat scar, telangiectasia, and/or whitening of the mucosa; 3) Absence of any palpable tumor or irregularity on digital rectal examination (DRE) and endoscopic ultrasonography (EUS); 4) If a biopsy is taken, it must be negative.
Time Frame: At Week 15
Population: FAS include all participants who are enrolled in the study and received at least 1 dose of study intervention.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Peposertib 50 mg + RT + Capecitabine: | Peposertib 100 mg + RT + Capecitabine: | Peposertib 150 mg + RT + Capecitabine: | Peposertib 250 mg + RT + Capecitabine:
Number analyzed (Participants) | 1 | 6 | 6 | 6
percentage of participants | 0.0 [0.0 to 97.5] | 16.7 [0.4 to 64.1] | 16.7 [0.4 to 64.1] | 16.7 [0.4 to 64.1]

10. Secondary Outcome: Time From Surgery to Local Recurrence
Description: Time from surgery to local recurrence defined as time from day of surgery to the date of the first documentation of progression of disease, flagged as local recurrence. Median time from surgery to local recurrence was estimated according to Kaplan-Meier method.
Time Frame: Time from surgery up to 15 months
Population: FAS include all participants who are enrolled in the study and received at least 1 dose of study intervention. Here, number of participants analyzed signifies those participants who underwent rectal surgery. As per the planned analysis, Kaplan-Meier estimates were planned to be presented overall, together with a summary of associated statistics (median survival time and survival rate estimates) including the corresponding 2-sided 95% Confidence Intervals (CIs) for this outcome measure.
Measure: Median (Full Range); unit: months
Groups:
- All Participants: Participants received peposertib 100 mg, 150 mg and 250 mg in their respective cohort once daily in combination with capecitabine 825 milligram per square meter (mg/m^2) twice daily 5 days per week and radiotherapy (RT) of 50 to 50.4 Gray (Gy) to the tumor area and 45 Gy to the electively irradiated tissues in 25 to 28 fractions up to 5.5 weeks treatment period.
Arm/Group | All Participants
Number analyzed (Participants) | 9
months | NA [2.8 to 15.0] — Due to small number of events, Median and CI could not be determined.

11. Secondary Outcome: Time From Surgery to Distant Metastasis
Description: Time from surgery to distant metastasis defined as time from day of surgery to the date of the first documentation of progression of disease, flagged as distant metastasis. Median time from surgery to distant metastasis was estimated according to Kaplan-Meier method.
Time Frame: Time from surgery up to 15 months
Population: FAS include all participants who are enrolled in the study and received at least 1 dose of study intervention. Here, number of participants analyzed signifies those participants who underwent rectal surgery. As per the planned analysis, Kaplan-Meier estimates were planned to be presented overall, together with a summary of associated statistics for this outcome measure.
Measure: Median (Full Range); unit: months
Arm/Group | All Participants
Number analyzed (Participants) | 9
months | NA [2.8 to 15.0] — Due to small number of events, Median and CI could not be determined.

12. Secondary Outcome: Neoadjuvant Rectal (NAR) Score
Description: The NAR formula includes the clinical tumor (cT) stage, pathologic tumor (pT), and node (pN) stage according to the tumor, node, metastasis classification system for colorectal cancers. The NAR formula is as follows:
  [5pN- 3 (cT- pT) + 12]2 / 9.61
  NAR score ranges from 0 to 100, whereas a score close to 100 is indicative of a poorer prognosis.
Time Frame: At Week 15
Population: FAS include all participants who are enrolled in the study and received at least 1 dose of study intervention. Here, "Number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peposertib 50 mg + RT + Capecitabine: | Peposertib 100 mg + RT + Capecitabine: | Peposertib 150 mg + RT + Capecitabine: | Peposertib 250 mg + RT + Capecitabine:
Number analyzed (Participants) | 0 | 2 | 2 | 5
score on a scale |  | 9.4 (7.95) | 13.8 (1.69) | 21.2 (12.11)

13. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Peposertib
Description: Cmax was obtained directly from the concentration versus time curve. One participant was assigned to receive peposertib 100 mg; however, this participant took peposertib 50 mg for FD 1 through FD 10 and then took peposertib 100 mg for remainder of study participation. PK results for this participant was summarized by actual dose received (50 mg) whereas non-PK results are summarized by planned dose (100 mg).
Time Frame: Pre-dose, 1, 2, 3, 4 and 6 hours post-dose on Fraction Day 1 and Fraction Day 9
Population: Pharmacokinetic (PK) analysis set included participants who received at least 1 dose of peposertib and have sufficient peposertib plasma concentration data to enable the calculation of at least 1 PK parameter. Sufficient concentration data is defined as at least 3 valid, post dose, concentration points in the PK profile to obtain any PK parameter.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Peposertib 50 mg + RT + Capecitabine: | Peposertib 100 mg + RT + Capecitabine: | Peposertib 150 mg + RT + Capecitabine: | Peposertib 250 mg + RT + Capecitabine:
Number analyzed (Participants) | 2 | 5 | 6 | 6
nanogram per milliliter (ng/mL)
  Fraction Day 1 | NA (NA) — Geometric mean and Geometric coefficient of variation was not estimable, if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation. | 593 (55.8) | 728 (24.1) | 1350 (55.5)
  Fraction Day 9 | NA (NA) — Geometric mean and Geometric coefficient of variation was not estimable, if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation. | 653 (50.4) | 792 (41.8) | 1760 (35.6)

14. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Last Sampling Time (Tlast) (AUC0-t) of Peposertib
Description: Area under the plasma concentration vs time curve from time zero to the last sampling time t at which the concentration was at or above the lower limit of quantification (LLQ). AUC0-t was to be calculated according to the mixed log-linear trapezoidal rule.
Time Frame: Pre-dose, 1, 2, 3, 4 and 6 hour post-dose on Fraction Day 1 and Fraction Day 9
Population: PK analysis set was used. One participant was assigned to receive peposertib 100 mg; however, this participant took peposertib 50 mg for FD 1 through FD 10 and then took peposertib 100 mg for remainder of study participation. PK results for this participant was summarized by actual dose received (50 mg) whereas non-PK results are summarized by planned dose (100 mg).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Peposertib 50 mg + RT + Capecitabine: | Peposertib 100 mg + RT + Capecitabine: | Peposertib 150 mg + RT + Capecitabine: | Peposertib 250 mg + RT + Capecitabine:
Number analyzed (Participants) | 2 | 5 | 6 | 6
hour*nanogram per milliliter (h*ng/mL)
  Fraction Day 1 | NA (NA) — Geometric mean and Geometric coefficient of variation was not estimable, if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation. | 2950 (69.8) | 4000 (33.3) | 7300 (71.7)
  Fraction Day 9: number analyzed (Participants) | 2 | 5 | 5 | 6
  Fraction Day 9 | NA (NA) — Geometric mean and Geometric coefficient of variation was not estimable, if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation. | 3450 (81.9) | 5540 (51.0) | 9450 (50.0)

15. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of Peposertib
Description: Time to reach the maximum plasma concentration (Tmax) was obtained directly from the concentration versus time curve.
Time Frame: Pre-dose, 1, 2, 3, 4 and 6 hour post-dose on Fraction Day 1 and Fraction Day 9
Population: as for outcome 14
Measure: Median (Full Range); unit: hours
Arm/Group | Peposertib 50 mg + RT + Capecitabine: | Peposertib 100 mg + RT + Capecitabine: | Peposertib 150 mg + RT + Capecitabine: | Peposertib 250 mg + RT + Capecitabine:
Number analyzed (Participants) | 2 | 5 | 6 | 6
hours
  Fraction Day 1 | NA [3.00 to 4.00] — As per plan analysis, it was planned to report only minimum and maximum values if number of participants analyzed was less than or equal to 2 (n ≤ 2). Only the number of non-missing observations, the minimum and maximum values had to be reported. | 1.00 [0.83 to 2.00] | 2.33 [1.07 to 2.97] | 2.43 [0.85 to 4.00]
  Fraction Day 9 | NA [2.00 to 3.22] — As per plan analysis, it was planned to report only minimum and maximum values if number of participants analyzed was less than or equal to 2 (n ≤ 2). Only the number of non-missing observations, the minimum and maximum values had to be reported. | 2.05 [0.83 to 2.25] | 2.09 [1.07 to 3.82] | 2.01 [0.92 to 7.33]

16. Secondary Outcome: Total Body Clearance Following Oral Administration (CL/f) of Peposertib
Description: The apparent total body clearance of study intervention following extravascular administration on FD1, taking into account the fraction of dose absorbed. CL/f = Dose oral (p.o.)/AUC0-inf. The predicted AUC0-inf should be used.
Time Frame: Pre-dose, 1, 2, 3, 4 and 6 hour post-dose on Fraction Day 1
Population: PK analysis set was used. One participant was assigned to receive peposertib 100 mg; however, this participant took peposertib 50 mg for FD 1 through FD 10 and then took peposertib 100 mg for remainder of study participation. PK results for this participant was summarized by actual dose received (50 mg) whereas non-PK results are summarized by planned dose (100 mg). Here, "Number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour
Arm/Group | Peposertib 50 mg + RT + Capecitabine: | Peposertib 100 mg + RT + Capecitabine: | Peposertib 150 mg + RT + Capecitabine: | Peposertib 250 mg + RT + Capecitabine:
Number analyzed (Participants) | 0 | 5 | 6 | 5
Liter per hour |  | 31.7 (74.5) | 34.5 (41.1) | 33.0 (87.6)

17. Secondary Outcome: Apparent Volume of Distribution (Vz/f) of Peposertib
Description: The apparent volume of distribution during the terminal phase following extravascular administration, based on the fraction of dose absorbed. Vz/f = Dose/(AUC0-inf multiplied by Lambda z) following single dose. Vz/f= Dose/(AUCtau*Lambda z) following multiple dose. One participant was assigned to receive peposertib 100 mg; however, this participant took peposertib 50 mg for FD 1 through FD 10 and then took peposertib 100 mg for remainder of study participation. PK results for this participant was summarized by actual dose received (50 mg) whereas non-PK results are summarized by planned dose (100 mg).
Time Frame: Pre-dose, 1, 2, 3, 4 and 6 hour post-dose on Fraction Day 1 and Fraction Day 9
Population: PK analysis set was used. Here, "Number of participants" analyzed signifies those participants who were evaluable for this outcome measure. Here, "Number Analyzed" signified those participants who were evaluable at specified timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Peposertib 50 mg + RT + Capecitabine: | Peposertib 100 mg + RT + Capecitabine: | Peposertib 150 mg + RT + Capecitabine: | Peposertib 250 mg + RT + Capecitabine:
Number analyzed (Participants) | 1 | 5 | 6 | 5
Liter
  Fraction Day 1: number analyzed (Participants) | 0 | 5 | 6 | 5
  Fraction Day 1 |  | 256 (60.3) | 274 (25.7) | 245 (64.1)
  Fraction Day 9: number analyzed (Participants) | 1 | 5 | 5 | 5
  Fraction Day 9 | NA (NA) — Geometric mean and Geometric coefficient of variation was not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation. | 261 (100.8) | 217 (43.7) | 234 (39.7)

18. Secondary Outcome: Apparent Terminal Half-life (t1/2) of Peposertib
Description: Terminal half-life is the time measured for the concentration to decrease by one half. Terminal half-life calculated by natural log 2 divided by lambda z. One participant was assigned to receive peposertib 100 mg; however, this participant took peposertib 50 mg for FD 1 through FD 10 and then took peposertib 100 mg for remainder of study participation. PK results for this participant was summarized by actual dose received (50 mg) whereas non-PK results are summarized by planned dose (100 mg).
Time Frame: Pre-dose, 1, 2, 3, 4 and 6 hour post-dose on Fraction Day 1 and Fraction Day 9
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Peposertib 50 mg + RT + Capecitabine: | Peposertib 100 mg + RT + Capecitabine: | Peposertib 150 mg + RT + Capecitabine: | Peposertib 250 mg + RT + Capecitabine:
Number analyzed (Participants) | 1 | 5 | 6 | 5
hours
  Fraction Day 1: number analyzed (Participants) | 0 | 5 | 6 | 5
  Fraction Day 1 |  | 5.60 (22.0) | 5.51 (29.0) | 5.14 (28.7)
  Fraction Day 9: number analyzed (Participants) | 1 | 5 | 5 | 5
  Fraction Day 9 | NA (NA) — Geometric mean and Geometric coefficient of variation was not estimable, if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation. | 6.28 (30.8) | 5.04 (61.0) | 6.12 (28.9)

ADVERSE EVENTS:
Time Frame: Baseline up to long term follow-up period (approximately Month 35)
Arm/Group | Peposertib 50 mg + RT + Capecitabine: | Peposertib 100 mg + RT + Capecitabine: | Peposertib 150 mg + RT + Capecitabine: | Peposertib 250 mg + RT + Capecitabine:
All-Cause Mortality (participants affected / at risk) | 0/1 | 1/6 | 1/6 | 1/6
Serious Adverse Events (participants affected / at risk) | 0/1 | 3/6 | 0/6 | 4/6
Other Adverse Events (participants affected / at risk) | 1/1 | 5/6 | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Peposertib 50 mg + RT + Capecitabine: (N=1) | Peposertib 100 mg + RT + Capecitabine: (N=6) | Peposertib 150 mg + RT + Capecitabine: (N=6) | Peposertib 250 mg + RT + Capecitabine: (N=6)
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0 | 2
Proctitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Peposertib 50 mg + RT + Capecitabine: (N=1) | Peposertib 100 mg + RT + Capecitabine: (N=6) | Peposertib 150 mg + RT + Capecitabine: (N=6) | Peposertib 250 mg + RT + Capecitabine: (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 4
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 2
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Anal incontinence (Gastrointestinal disorders) | 0 | 1 | 2 | 0
Anal inflammation (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 5 | 3 | 5
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dyschezia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 4 | 2 | 2
Proctalgia (Gastrointestinal disorders) | 0 | 3 | 3 | 1
Proctitis (Gastrointestinal disorders) | 1 | 2 | 2 | 3
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 2 | 3
Rectal tenesmus (Gastrointestinal disorders) | 0 | 0 | 2 | 5
Rectal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 3
Fatigue (General disorders) | 1 | 5 | 3 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0
Secretion discharge (General disorders) | 0 | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 1
Vaginal infection (Infections and infestations) | 0 | 0 | 0 | 1
Anal injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Radiation skin injury (Injury, poisoning and procedural complications) | 1 | 3 | 2 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 2 | 2 | 3
Platelet count decreased (Investigations) | 0 | 1 | 0 | 1
Weight decreased (Investigations) | 0 | 1 | 2 | 0
White blood cell count decreased (Investigations) | 0 | 2 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 3 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 3 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
Dizziness postural (Nervous system disorders) | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 1
Personality change (Psychiatric disorders) | 1 | 0 | 0 | 0
Bladder spasm (Renal and urinary disorders) | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 1 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urinary hesitation (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0
Peripheral embolism (Vascular disorders) | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
As decided by sponsor study was discontinued prior to the initiation of the Phase II part of the study; therefore, results only from the Phase Ib part of the study was reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-05-06): https://cdn.clinicaltrials.gov/large-docs/89/NCT03770689/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-07): https://cdn.clinicaltrials.gov/large-docs/89/NCT03770689/SAP_001.pdf